CLINICAL TRIAL: NCT06295276
Title: Does a Teletherapy-guided Exercise Programme Improve Pain Intensity, Disability, and Quality of Life in Nursing Students With Back and Neck Pain Compared to a Control Group?
Brief Title: Effect of Teletherapy-supported Training on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hochschule Osnabruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSOsnabruck
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Neck Pain
Keywords: teletherapy
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: Parallel comparative randomized controlled trial
Masking Description: Allocation concealment:
  The results of the allocation sequence are placed in sequentially numbered, opaque, and sealed envelopes by an independent researcher to ensure confidentiality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): a six-week muscle training program with 5 exercises 3 times a week as video-guided exercises for homework alone and the same exercises once a week guided by Zoom. The program lasts 6 weeks
  Interventions: Other: teletherapy-guided exercise programme
- Waiting list/control intervention/delayed teletherapy intervention (Other): After the 6 weeks, participants are offered the opportunity to take part in the intervention program (see above)
  Interventions: Other: Waiting list/control intervention/delayed teletherapy intervention

INTERVENTIONS:
Other: teletherapy-guided exercise programme — Exercise program guided by online sessions. Subjects perform this exercise program three times a week at home, so that they complete four sessions per week for six weeks. The duration of a session is approximately twenty minutes. There are six exercises with three sets and about fifteen repetitions. Subjects in the treatment group also receive an instructional video. The subjects keep a diary in which they record their adherence to the treatment protocol at home.
  At the beginning of the intervention and after the sixth week, participants are assessed with ODI, NDI and SF36-Short and NRS-11 scales. At the end, we use the Global Rating Scale.
  Arms: Intervention
Other: Waiting list/control intervention/delayed teletherapy intervention — Subjects in the control group will be advised to maintain their daily routine but will be asked to refrain from other treatments to avoid co-interventions during the 6-week study period. However, the use of painkillers such as non-steroidal anti-inflammatory analgesics (NSAIDs) taken by study participants in all groups for more than 3 months is allowed and will be documented (taking a pragmatic approach). Any change in medication will be monitored and documented by the PT at each visit.
  Arms: Waiting list/control intervention/delayed teletherapy intervention

SUMMARY:
Design: This study is a pilot randomized controlled trial (RCT) with two-arm parallel groups, the gold standard for determining treatment efficacy. The flowchart (see appendix) provides an overview of the study design. Participants are randomized and stratified by age into intervention group and waiting list group.

The intervention is teletherapy-supported muscular training for 20 minutes 4 times a week.

The duration of the intervention is six weeks in total. At the beginning Neck Disability Index (NDI), Oswestry Disability Index (ODI), Short-Form-36 (SF36), and the Numerical rating Scale (NRS) are collected. After six weeks, the same outcome measures and the global rating scale

DETAILED DESCRIPTION:
Intervention of interest: As already mentioned, the protocol of interest is an exercise program supported by online sessions (teletherapy). Exercise routines related to the individual areas of the spine as a functional unit were created based on evidence-based conclusions, especially considering muscle chain activity and appropriate loading parameters

The teletherapy exercise program is carried out once a week via ZOOM by a physiotherapist with thirty years of experience in treating patients with musculoskeletal disorders. Participants are also encouraged to carry out this exercise program themselves at home three times a week so that they have four sessions per week for six weeks. The duration of each session is approximately twenty minutes per session. There are six exercises with three sets and about fifteen repetitions within thirty seconds per set. Exercise description with rationale for exercise selection"). Subjects in the treatment group will also receive a video, rhythm and music files and written materials to help them follow the exercise routines at home, as well as a rubber band. Subjects are also asked to keep a diary in which they record their adherence to the home treatment protocol.

At the beginning of the intervention and after the seventh week, the participants are each assessed with the Patient Reported Outcomes (PROMs), namely ODI, NDI and SF36 short and NRS 11-point scales. At the end of the intervention, participants are interviewed using the Global Rating Scale. Below is a brief description of these instruments.

Control group:

Subjects in the control group will be advised to maintain their daily routine but will be asked to refrain from other treatments such as physical Therapy (PT), osteopathy, chiropractic as well as other therapeutic exercise (TE) therapies to avoid co-interventions during the 6-week study period. However, pain medication taken by study participants for more than 3 months in all groups, such as non-steroidal anti-inflammatory analgesics (NSAIDs), will be permitted and documented (taking a pragmatic approach). Any change in medication will be monitored and recorded by the PT at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students between 18 and 60 years of any gender
* Self-reported chronic neck and back pain in the last six months (more than three months as described by the International Association for the Study of Pain (IASP)).
* Speak and understand German

Exclusion Criteria:

Surgery in the last year on the spine, cervical, thoracic, or lumbar spine

* Currently on sick leave
* Acute back pain
* Severe neurological injuries or symptoms
* Acute trauma to the musculoskeletal system
* Renal insufficiency, dialysis
* Severe impairment of the ability to grip with the hand, e.g., rheumatoid arthritis.
* Severe cardiovascular diseases, e.g. heart failure
* Severe respiratory diseases, e.g., Chronic Obstructive Pulmonary Disease-COPD
* Nystagmus
* Falling tendency/balance disorders
* Latex allergy, as rubber band may be made of latex
* Lack of ability to stand, inability to stand safely without the help of a person or object.
* A spine-specific pain therapy drug treatment within the last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Baseline-6 weeks
  10 questions with possible answers ranging from "no pain" to "the worst pain you can imagine", questions for pain intensity, personal hygiene, lifting, reading, headaches, concentration, work, driving, sleeping and the last item leisure activities and recreation.
  Rating:
  Mild complaints 0 points, the most severe complaints with a maximum of 5 points. Maximum score 50 points.
  Score is divided by the possible total score. This value is multiplied by 100% to obtain the score. o (Current restriction : 50) X 100% = score in the NDI <=8% mild symptoms. >40 has very severe symptoms
Oswestry Disability Index (ODI) | Baseline-6 weeks
  Extent of pain-related functional limitations in people with back pain. 10 questions with six possible answers each: Pain intensity, self-care, lifting, walking, sitting or standing, sleeping, sex life, social life and traveling.
  Answer options range from "no restrictions due to pain" to "greatest perceived restriction of an activity due to pain".
  Evaluation:
  Points achieved ( )/max. points (50) x100 = % Interpretation: 0% = no restriction, 100% = max. restriction.
NRS Numeric rating scale for pain | Baseline- 6 weeks
  The Numerical Rating Scale for Pain (NRS) is usually between 0 and 10, with 0 being "no pain" and 10 being "the worst pain imaginable" In a numerical rating scale question, respondents are asked to rate their perceived pain on a predetermined numerical scale. The scale is an ordered number scale with a fixed range that represents the extremes of the measured value

SECONDARY OUTCOMES:
Short-Form: SF 36-Quality of life | Baseline- 6 weeks
  SF 36-Quality of life he SF-36 questionnaire (Short Form Health 36) is a questionnaire on quality of life.
  For information on the general. 8 different dimensions Vitality - Physical functioning - Physical pain - General health perception - Physical role functioning - Emotional role functioning - Social role functioning - Psychological well-being For the evaluation, all answers are first converted into predefined points with the help of an evaluation key. The average value of all questions of the respective health dimension
Global rating scale | 6 weeks
  The Global Rating Scale (GRS) is described as a useful measurement tool with the aim of assessing clinical competence at a general level based on specific word dimensions, measuring instrument to determine the effect of the intervention . This scale is used by us in the study to assess the changes experienced by the patient as a result of treatments or other interventions. Our subjects are asked to rate the change they have experienced after treatment for neck pain and low back pain (LBP) pain using a Global Rating Scale (GRS). Therefore, this questionnaire is only used for the final measurement.
  Participants rate their state of health now compared to before the intervention.
  The values range from -7 to 7. It is measured with -7 as "very much worse", 0 as "unchanged" and 7 as the maximum best value "very much better".

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonie Pflege Schule, Osnabrück, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adorno ML, Brasil-Neto JP. Assessment of the quality of life through the SF-36 questionnaire in patients with chronic nonspecific low back pain. Acta Ortop Bras. 2013 Jul;21(4):202-7. doi: 10.1590/S1413-78522013000400004. PMID 24453669
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Bremer A, Andersson Hagiwara M, Tavares W, Paakkonen H, Nystrom P, Andersson H. Translation and further validation of a global rating scale for the assessment of clinical competence in prehospital emergency care. Nurse Educ Pract. 2020 Aug;47:102841. doi: 10.1016/j.nepr.2020.102841. Epub 2020 Jul 16. PMID 32768897
- [Background] Buskard ANL, Jacobs KA, Eltoukhy MM, Strand KL, Villanueva L, Desai PP, Signorile JF. Optimal Approach to Load Progressions during Strength Training in Older Adults. Med Sci Sports Exerc. 2019 Nov;51(11):2224-2233. doi: 10.1249/MSS.0000000000002038. PMID 31107348
- [Background] Young BA, Walker MJ, Strunce JB, Boyles RE, Whitman JM, Childs JD. Responsiveness of the Neck Disability Index in patients with mechanical neck disorders. Spine J. 2009 Oct;9(10):802-8. doi: 10.1016/j.spinee.2009.06.002. Epub 2009 Jul 25. PMID 19632904
- [Background] Quentin C, Bagheri R, Ugbolue UC, Coudeyre E, Pelissier C, Descatha A, Menini T, Bouillon-Minois JB, Dutheil F. Effect of Home Exercise Training in Patients with Nonspecific Low-Back Pain: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Aug 10;18(16):8430. doi: 10.3390/ijerph18168430. PMID 34444189
- [Background] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937
- [Background] Dal Farra F, Arippa F, Arru M, Cocco M, Porcu E, Tramontano M, Monticone M. Effects of exercise on balance in patients with non-specific low back pain: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2022 Jun;58(3):423-434. doi: 10.23736/S1973-9087.21.07293-2. Epub 2021 Oct 12. PMID 34636528
- [Background] Eckard T, Lopez J, Kaus A, Aden J. Home exercise program compliance of service members in the deployed environment: an observational cohort study. Mil Med. 2015 Feb;180(2):186-91. doi: 10.7205/MILMED-D-14-00306. PMID 25643386
- [Background] Ennis S, McGregor G, Hamborg T, Jones H, Shave R, Singh SJ, Banerjee P. Randomised feasibility trial into the effects of low-frequency electrical muscle stimulation in advanced heart failure patients. BMJ Open. 2017 Aug 11;7(8):e016148. doi: 10.1136/bmjopen-2017-016148. PMID 28801415
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Filho RAA, Oliveira JJG, Zovico PVC, Rica RL, Barbosa WA, Machado AF, Evangelista AL, Costa EC, Bergamin M, Baker JS, Bocalini DS. Effects of music on psychophysiological responses during high intensity interval training using body weight exercises. Physiol Behav. 2022 Oct 15;255:113931. doi: 10.1016/j.physbeh.2022.113931. Epub 2022 Jul 28. PMID 35907471
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Gloth MJ, Matesi AM. Physical therapy and exercise in pain management. Clin Geriatr Med. 2001 Aug;17(3):525-35, vii. doi: 10.1016/s0749-0690(05)70084-7. PMID 11459719
- [Background] Grotle M, Garratt AM, Krogstad Jenssen H, Stuge B. Reliability and construct validity of self-report questionnaires for patients with pelvic girdle pain. Phys Ther. 2012 Jan;92(1):111-23. doi: 10.2522/ptj.20110076. Epub 2011 Oct 20. PMID 22016375
- [Background] Helms ER, Cronin J, Storey A, Zourdos MC. Application of the Repetitions in Reserve-Based Rating of Perceived Exertion Scale for Resistance Training. Strength Cond J. 2016 Aug;38(4):42-49. doi: 10.1519/SSC.0000000000000218. Epub 2016 Aug 3. PMID 27531969
- [Background] Herr KA, Spratt K, Mobily PR, Richardson G. Pain intensity assessment in older adults: use of experimental pain to compare psychometric properties and usability of selected pain scales with younger adults. Clin J Pain. 2004 Jul-Aug;20(4):207-19. doi: 10.1097/00002508-200407000-00002. PMID 15218405
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Javdaneh N, Ambrozy T, Barati AH, Mozafaripour E, Rydzik L. Focus on the Scapular Region in the Rehabilitation of Chronic Neck Pain Is Effective in Improving the Symptoms: A Randomized Controlled Trial. J Clin Med. 2021 Aug 8;10(16):3495. doi: 10.3390/jcm10163495. PMID 34441791
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Jorritsma W, Dijkstra PU, de Vries GE, Geertzen JH, Reneman MF. Detecting relevant changes and responsiveness of Neck Pain and Disability Scale and Neck Disability Index. Eur Spine J. 2012 Dec;21(12):2550-7. doi: 10.1007/s00586-012-2407-8. Epub 2012 Jul 3. PMID 22752592
- [Background] Jorritsma W, de Vries GE, Dijkstra PU, Geertzen JH, Reneman MF. Neck Pain and Disability Scale and Neck Disability Index: validity of Dutch language versions. Eur Spine J. 2012 Jan;21(1):93-100. doi: 10.1007/s00586-011-1920-5. Epub 2011 Aug 4. PMID 21814745
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Kang T, Kim B. Cervical and scapula-focused resistance exercise program versus trapezius massage in patients with chronic neck pain: A randomized controlled trial. Medicine (Baltimore). 2022 Sep 30;101(39):e30887. doi: 10.1097/MD.0000000000030887. PMID 36181044
- [Background] Kendrick DB, Strout TD. The minimum clinically significant difference in patient-assigned numeric scores for pain. Am J Emerg Med. 2005 Nov;23(7):828-32. doi: 10.1016/j.ajem.2005.07.009. PMID 16291435
- [Background] Letafatkar A, Rabiei P, Alamooti G, Bertozzi L, Farivar N, Afshari M. Effect of therapeutic exercise routine on pain, disability, posture, and health status in dentists with chronic neck pain: a randomized controlled trial. Int Arch Occup Environ Health. 2020 Apr;93(3):281-290. doi: 10.1007/s00420-019-01480-x. Epub 2019 Oct 25. PMID 31654125
- [Background] Lin G, Zhao X, Wang W, Wilkinson T. The relationship between forward head posture, postural control and gait: A systematic review. Gait Posture. 2022 Oct;98:316-329. doi: 10.1016/j.gaitpost.2022.10.008. Epub 2022 Oct 14. PMID 36274469
- [Background] Duenas L, Aguilar-Rodriguez M, Voogt L, Lluch E, Struyf F, Mertens MGCAM, Meulemeester K, Meeus M. Specific versus Non-Specific Exercises for Chronic Neck or Shoulder Pain: A Systematic Review. J Clin Med. 2021 Dec 18;10(24):5946. doi: 10.3390/jcm10245946. PMID 34945241
- [Background] McCarthy MJ, Grevitt MP, Silcocks P, Hobbs G. The reliability of the Vernon and Mior neck disability index, and its validity compared with the short form-36 health survey questionnaire. Eur Spine J. 2007 Dec;16(12):2111-7. doi: 10.1007/s00586-007-0503-y. Epub 2007 Oct 6. PMID 17922152
- [Background] Mueller J, Niederer D. Dose-response-relationship of stabilisation exercises in patients with chronic non-specific low back pain: a systematic review with meta-regression. Sci Rep. 2020 Oct 9;10(1):16921. doi: 10.1038/s41598-020-73954-9. PMID 33037280
- [Background] Naugle KM, Fillingim RB, Riley JL 3rd. A meta-analytic review of the hypoalgesic effects of exercise. J Pain. 2012 Dec;13(12):1139-50. doi: 10.1016/j.jpain.2012.09.006. Epub 2012 Nov 8. PMID 23141188
- [Background] Ogura K, Bartelstein MK, Yakoub MA, Nikolic Z, Boland PJ, Healey JH. Minimal clinically important differences in SF-36 global score: Current value in orthopedic oncology. J Orthop Res. 2021 Oct;39(10):2116-2123. doi: 10.1002/jor.24944. Epub 2020 Dec 20. PMID 33617087
- [Background] Ogura K, Yakoub MA, Christ AB, Fujiwara T, Nikolic Z, Boland PJ, Healey JH. What Are the Minimum Clinically Important Differences in SF-36 Scores in Patients with Orthopaedic Oncologic Conditions? Clin Orthop Relat Res. 2020 Sep;478(9):2148-2158. doi: 10.1097/CORR.0000000000001341. PMID 32568896
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] Polaski AM, Phelps AL, Kostek MC, Szucs KA, Kolber BJ. Exercise-induced hypoalgesia: A meta-analysis of exercise dosing for the treatment of chronic pain. PLoS One. 2019 Jan 9;14(1):e0210418. doi: 10.1371/journal.pone.0210418. eCollection 2019. PMID 30625201
- [Background] Pool JJ, Ostelo RW, Hoving JL, Bouter LM, de Vet HC. Minimal clinically important change of the Neck Disability Index and the Numerical Rating Scale for patients with neck pain. Spine (Phila Pa 1976). 2007 Dec 15;32(26):3047-51. doi: 10.1097/BRS.0b013e31815cf75b. PMID 18091500
- [Background] Reppa CM, Bogdanis GC, Stavrou NAM, Psychountaki M. The Effect of Aerobic Fitness on Psychological, Attentional and Physiological Responses during a Tabata High-Intensity Interval Training Session in Healthy Young Women. Int J Environ Res Public Health. 2023 Jan 5;20(2):1005. doi: 10.3390/ijerph20021005. PMID 36673761
- [Background] Rice D, Nijs J, Kosek E, Wideman T, Hasenbring MI, Koltyn K, Graven-Nielsen T, Polli A. Exercise-Induced Hypoalgesia in Pain-Free and Chronic Pain Populations: State of the Art and Future Directions. J Pain. 2019 Nov;20(11):1249-1266. doi: 10.1016/j.jpain.2019.03.005. Epub 2019 Mar 21. PMID 30904519
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Saltychev M, Mattie R, McCormick Z, Barlund E, Laimi K. Psychometric properties of the Oswestry Disability Index. Int J Rehabil Res. 2017 Sep;40(3):202-208. doi: 10.1097/MRR.0000000000000226. PMID 28368870
- [Background] Saltychev M, Vastamaki H, Mattie R, McCormick Z, Vastamaki M, Laimi K. Psychometric Properties of the Pain Numeric Rating Scale When Applied to Multiple Body Regions among Professional Musicians. PLoS One. 2016 Sep 7;11(9):e0161874. doi: 10.1371/journal.pone.0161874. eCollection 2016. PMID 27603011
- [Background] Schellingerhout JM, Verhagen AP, Heymans MW, Koes BW, de Vet HC, Terwee CB. Measurement properties of disease-specific questionnaires in patients with neck pain: a systematic review. Qual Life Res. 2012 May;21(4):659-70. doi: 10.1007/s11136-011-9965-9. Epub 2011 Jul 7. PMID 21735306
- [Background] Sheahan PJ, Nelson-Wong EJ, Fischer SL. A review of culturally adapted versions of the Oswestry Disability Index: the adaptation process, construct validity, test-retest reliability and internal consistency. Disabil Rehabil. 2015;37(25):2367-74. doi: 10.3109/09638288.2015.1019647. Epub 2015 Mar 4. PMID 25738913
- [Background] Steffen T, Seney M. Test-retest reliability and minimal detectable change on balance and ambulation tests, the 36-item short-form health survey, and the unified Parkinson disease rating scale in people with parkinsonism. Phys Ther. 2008 Jun;88(6):733-46. doi: 10.2522/ptj.20070214. Epub 2008 Mar 20. Erratum In: Phys Ther. 2010 Mar;90(3):462. PMID 18356292
- [Background] Sutanto D, Ho RST, Poon ETC, Yang Y, Wong SHS. Effects of Different Trunk Training Methods for Chronic Low Back Pain: A Meta-Analysis. Int J Environ Res Public Health. 2022 Mar 1;19(5):2863. doi: 10.3390/ijerph19052863. PMID 35270557
- [Background] Tataryn N, Simas V, Catterall T, Furness J, Keogh JWL. Posterior-Chain Resistance Training Compared to General Exercise and Walking Programmes for the Treatment of Chronic Low Back Pain in the General Population: A Systematic Review and Meta-Analysis. Sports Med Open. 2021 Mar 8;7(1):17. doi: 10.1186/s40798-021-00306-w. PMID 33683497
- [Background] Vaegter HB, Handberg G, Graven-Nielsen T. Similarities between exercise-induced hypoalgesia and conditioned pain modulation in humans. Pain. 2014 Jan;155(1):158-167. doi: 10.1016/j.pain.2013.09.023. Epub 2013 Sep 26. PMID 24076045
- [Background] Verbrugghe J, Agten A, Stevens S, Hansen D, Demoulin C, O Eijnde B, Vandenabeele F, Timmermans A. Exercise Intensity Matters in Chronic Nonspecific Low Back Pain Rehabilitation. Med Sci Sports Exerc. 2019 Dec;51(12):2434-2442. doi: 10.1249/MSS.0000000000002078. PMID 31269004
- [Background] Verbrugghe J, Agten A, Stevens S, Vandenabeele F, Roussel N, Verbunt J, Goossens N, Timmermans A. High intensity training improves symptoms of central sensitization at six-month follow-up in persons with chronic nonspecific low back pain: Secondary analysis of a randomized controlled trial. Braz J Phys Ther. 2023 Mar-Apr;27(2):100496. doi: 10.1016/j.bjpt.2023.100496. Epub 2023 Mar 17. PMID 36963161
- [Background] Verhagen AP. Physiotherapy management of neck pain. J Physiother. 2021 Jan;67(1):5-11. doi: 10.1016/j.jphys.2020.12.005. Epub 2020 Dec 24. No abstract available. PMID 33358545
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Whitehead AL, Sully BG, Campbell MJ. Pilot and feasibility studies: is there a difference from each other and from a randomised controlled trial? Contemp Clin Trials. 2014 May;38(1):130-3. doi: 10.1016/j.cct.2014.04.001. Epub 2014 Apr 13. PMID 24735841
- [Background] Wilhelm MP, Donaldson M, Griswold D, Learman KE, Garcia AN, Learman SM, Cleland JA. The Effects of Exercise Dosage on Neck-Related Pain and Disability: A Systematic Review With Meta-analysis. J Orthop Sports Phys Ther. 2020 Nov;50(11):607-621. doi: 10.2519/jospt.2020.9155. PMID 33131392
- [Background] Yasa ME, Un Yildirim N, Demir P. The effects of a 6-Week balance training in addition to conventional physiotherapy on pain, postural control, and balance confidence in patients with cervical disc herniation: a randomized controlled trial. Somatosens Mot Res. 2021 Mar;38(1):60-67. doi: 10.1080/08990220.2020.1845136. Epub 2020 Nov 10. PMID 33172321
- [Background] Yildiz TI, Turgut E, Duzgun I. Neck and Scapula-Focused Exercise Training on Patients With Nonspecific Neck Pain: A Randomized Controlled Trial. J Sport Rehabil. 2018 Sep 1;27(5):403-412. doi: 10.1123/jsr.2017-0024. Epub 2018 Jul 25. PMID 28605288
- [Background] de Zoete RM, Armfield NR, McAuley JH, Chen K, Sterling M. Comparative effectiveness of physical exercise interventions for chronic non-specific neck pain: a systematic review with network meta-analysis of 40 randomised controlled trials. Br J Sports Med. 2020 Nov 2:bjsports-2020-102664. doi: 10.1136/bjsports-2020-102664. Online ahead of print. PMID 33139256
- [Background] Zourdos MC, Klemp A, Dolan C, Quiles JM, Schau KA, Jo E, Helms E, Esgro B, Duncan S, Garcia Merino S, Blanco R. Novel Resistance Training-Specific Rating of Perceived Exertion Scale Measuring Repetitions in Reserve. J Strength Cond Res. 2016 Jan;30(1):267-75. doi: 10.1519/JSC.0000000000001049. PMID 26049792
- [Background] Hrvatin, I./Puh, U. (2000). Measurement properties of the numerical pain rating scale. Patients with musculoskeletal impairment of the limbs. Slovenian Medical Journal, 1-9. https://doi.org/10.6016/ZdravVestn.3108.
- [Background] Iohom, G. (2006). Clinical Assessment of Postoperative Pain. Postoperative Pain Management, 102. Available online at DOI:10.1016/B978-1-4160-2454-5.50016-3.
- See also: Appendices_additional_information — https://drive.google.com/file/d/1pjgPQwPqNod6kXGwLzJg2Tys2hdWb_Pv/view?usp=drive_link